CLINICAL TRIAL: NCT07296679
Title: The Effect of Hand Massage on Anxiety and Comfort of Bariatric Surgery Patients: A Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Dilek Güneş, Associate Professor, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FiratOU
Record Dates: First submitted 2025-11-25; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Hand Massage; Anxiety
Keywords: Hand massage; anxiety; comfort; nursing
MeSH Terms: conditions — Anxiety Disorders | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: This randomised controlled experimental study
Who Masked: Participant
Masking Description: Single (Participant) By drawing lots, the first set was chosen to correspond to the experimental group and the second set to correspond to the control group for the two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Upon admission to the General Surgery clinic, patients were apprised of the study's objective, and their written and verbal agreement was acquired. Prior to the preoperative hand massage, the Patient Information Form, State-Trait Anxiety Inventory (STAI), and Short Form General Comfort Questionnaire (SGCQ) were administered to the patients in the general surgery clinic's patient room via face-to-face interviews.
  The patient rooms were single-occupancy, naturally lit, windowed, calm, quiet, and located within the clinic. Immediately before surgery, classic massage techniques including petrissage, friction, and kneading were applied to both hands for 10 minutes using baby oil on the palms, backs of the hands, and fingers. The hand massage was performed while the patient was in bed. The application lasted approximately 25 minutes. After the hand massage, State-Trait Anxiety Inventory (STAI) and General Comfort Scale-Short Form (SGCQ) were administered to the patients as post-test.
  Interventions: Other: Experimental Group
- Control group (No Intervention): No intervention other than the clinic protocol was applied to this group. In the control group, Patient Information Form, State-Trait Anxiety Inventory (STAI), General Comfort Scale-Short Form (SGCQ) were administered as pre-test before the operation. Just before the operation, State-Trait Anxiety Inventory (STAI) and General Comfort Scale-Short Form were administered as post-test.

INTERVENTIONS:
Other: Experimental Group — Upon admission to the General Surgery clinic, patients were apprised of the study's objective, and their written and verbal agreement was acquired. Prior to the preoperative hand massage, the Patient Information Form, State-Trait Anxiety Inventory (STAI), and Short Form General Comfort Questionnaire (SGCQ) were administered to the patients in the general surgery clinic's patient room via face-to-face interviews. The patient rooms were single-occupancy, naturally lit, windowed, calm, quiet, and located within the clinic. Immediately before surgery, classic massage techniques including petrissage, friction, and kneading were applied to both hands for 10 minutes using baby oil on the palms, backs of the hands, and fingers. The hand massage was performed while the patient was in bed. The application lasted approximately 25 minutes. After the hand massage, State-Trait Anxiety Inventory (STAI) and General Comfort Scale-Short Form (SGCQ) were administered to the patients as post-test.
  Other Names: Procedure/Surgery
  Arms: Experimental group

SUMMARY:
This study was conducted to determine the effect of hand massage on anxiety and comfort levels in bariatric surgery patients.

DETAILED DESCRIPTION:
This study was conducted to determine the effect of hand massage on anxiety and comfort levels in bariatric surgery patients. This randomised controlled trial was conducted in the General Surgery Clinic of a University Hospital in eastern Turkey with all adult patients undergoing bariatric surgery between September 2024 - March 2025. The sample consisted of 90 randomised patients who received hand massage and received only routine care. Data were collected using the Patient Information Form, State-Trait Anxiety Inventory (STAI), General Comfort Scale-Short Form (SGCQ).

ELIGIBILITY:
Inclusion criteria:

* Aged 18 or older
* Not having a speech problem or hearing loss
* Not having any condition that would reduce comprehension and understanding abilities
* Agreeing to participate in the study
* Having a body mass index (BMI) ≥ 30.

Exclusion criteria:

* Having compromised tissue and skin on the forearm or hands (e.g., wounds, eczema, inflammation, phlebitis, arthritis, and rashes)
* Having an intravenous catheter in the back of the hand.

Ages: 35 Years to 53 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2024-04-14 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
State Anxiety Inventory (STAI) | two weeks
  The scale was developed by Spielberger et al. Reliability and validity were carried out by Öner and Le Compte. The scale consists of two sub-units that measure anxiety separately, but in this study, the state anxiety scale that the individual feels indirectly from the stressful situation will be used. It is a 4-point Likert-type scale consisting of 20 items and short statements. The total score obtained from the scale varies between 20 and 80, and a high score indicates a high level of anxiety.

SECONDARY OUTCOMES:
General Comfort Scale-Short Form (SGCQ) | two weeks
  It was developed by Kolcaba to determine the comfort requirements of the individual. The Turkish validity and reliability study of the scale was conducted by Sarıtaş et al. In the evaluation of the scale, negative items (items 2, 3, 7, 9, 11, 18, 20, 21, 23, 24, 27) are reverse coded and summed. This 6-point Likert-type scale consisting of 28 items consists of three sub-dimensions: refreshment (1-9 items), relaxation (10-18 items) and superiority (19-28 items). The lowest score that can be obtained from the scale is 28 and the highest score is 168. As the score obtained from the scale decreases, it indicates that the comfort level of the individual is low.

CONTACTS AND LOCATIONS:
Overall Officials: DİLEK GÜNEŞ, Principal Investigator — FIRAT ÜNİVERSİTESİ
Locations (1):
- Firat Universty, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No